CLINICAL TRIAL: NCT06417606
Title: A Single-arm, Prospective Clinical Study of Lenvatinib and Adebrelimab Combined With GEMOX in the Perioperative Treatment of Potentially Resectable Intrahepatic Cholangiocarcinoma
Brief Title: Lenvatinib and Adebrelimab Combined With GEMOX in the Perioperative Treatment of Potentially Resectable Intrahepatic Cholangiocarcinoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhiyong Huang (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEC-ZN-01-AF 09
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib and Adebrelimab Combined With GEMOX（Gemcitabine and oxaliplatin） (Experimental): Lenvatinib（oral，12mg once daily if body weight ≥60Kg; Body weight < 60Kg, 8mg/ day）； Adebrelimab（intravenous drip，1200mg once every 3 weeks）； GEMOX（intravenous drip，Gemcitabine 1000mg/m2, 2 times every 3 weeks d1+d8; intravenous drip，Oxaliplatin, 100mg/m2, was given every 3 weeks）
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib（oral，12mg once daily if body weight ≥60Kg; Body weight < 60Kg, 8mg/ day）； Adebrelimab（intravenous drip，1200mg once every 3 weeks）； GEMOX（intravenous drip，Gemcitabine 1000mg/m2, 2 times every 3 weeks d1+d8; intravenous drip，Oxaliplatin, 100mg/m2, was given every 3 weeks）
  Other Names: Adebrelimab; GEMOX（Gemcitabine and oxaliplatin）

SUMMARY:
A single-arm, prospective clinical study was conducted to enroll 20 subjects. Each subject was treated with oral Lenvatinib + Adebrelimab + GEMOX (gemcitabine + oxaliplatin). The treatment phase before surgery was 3 cycles, and the evaluation was performed every 2 cycles. The evaluation was repeated before surgery, and the decision of surgery was made according to the evaluation results.

To evaluate the efficacy and safety of Lenvatinib and Adebrelimab combined with GEMOX in the perioperative treatment of potentially resectable intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participated in this study, signed informed consent, aged 18-80 years
* Patients with locally advanced intrahepatic cholangiocarcinoma: (meet at least one of the following) A, the number of intrahepatic tumors was 2-3 B, the intrahepatic tumor is single but >5cm in diameter C, the tumor was close to the 1/2 grade branch of the hepatic pedicle, making RO resection difficult D. Lymph node metastasis: MRI or PET/CT suggested regional lymph node metastasis
* The WHO/ECOG PS score was 0-1
* Imaging examination (CT/MRI/PET-CT) showed no distant metastasis
* Child-Pugh grade: A (≤6 points)
* Expected survival time ≥6 months
* No previous systemic treatment for hepatocellular carcinoma, including chemotherapy, targeted therapy, immunotherapy, etc. Patients who had undergone previous curative surgery or curative ablation were allowed, except those who had a recurrence within 2 years after curative surgery and those who had received other previous local treatment
* If you have hepatitis B virus (HBV) infection, such as HBsAg positive, you need to test HBV-DNA, and HBV-DNA should be less than 500IU/mL (; Patients with HBV-DNA of more than 500 IU per milliliter received antiviral therapy (only nucleoside agents such as entecavir, tenofovir dipivoxil fumarate, and tenofovir propofol fumarate tablets) for at least 1 week before randomization and had a decrease in viral copy number by a factor of more than 10. For patients with HBV infection, antiviral therapy should be received throughout the study period. Patients who are positive for hepatitis C virus (HCV) -RNA must receive antiviral therapy according to treatment guidelines
* Organs and bone marrow are sufficiently functional, defined as follows:

  1. hemoglobin ≥9g/dL
  2. absolute neutrophil count ≥1.5 × 109/L
  3. platelet count ≥ 100 × 109/L
  4. serum bilirubin ≤2.0× upper limit of normal (ULN); This condition does not apply to patients with proven Gilbert's syndrome. Any clinically significant biliary obstruction had to be relieved prior to enrollment in the study.
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be ≤2.5×ULN. For patients with liver metastases, ALT and AST should be ≤5 × ULN.

Exclusion Criteria:

* The investigator deemed the subject unfit to participate in the study
* Have active autoimmune disease or a history of autoimmune disease with possible recurrence (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism)
* Use of immunosuppressant or systemic hormone therapy to achieve immunosuppression within 2 weeks before treatment (dose >10mg/ day of prednisone or other effective hormones)
* patients with active infection, unexplained fever ≥38.5℃ within 1 week before randomization, or white blood cell count >15×109/L during screening; Therapeutic antibiotics, administered orally or intravenously, were given within 2 weeks before randomization
* Patients with innate or acquired immune deficiency (e.g., HIV infection)
* History of other primary malignancies, with the exception of malignancies treated with curative treatment, known absence of active disease ≥5 years before the first study intervention, and low potential risk of recurrence; Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or lentigo maligna that has received potentially curative treatment; Or carcinoma in situ that has been adequately treated without evidence of disease
* Patients with clinically significant bleeding symptoms or a clear bleeding tendency within 6 months before treatment, such as gastrointestinal bleeding, severe esophagogastric varices, hemorrhagic gastric ulcer, or angiitis, can be reexamined if fecal occult blood is positive at baseline, and if it is still positive after reexamination, gastroscopy is required
* Known inherited or acquired bleeding (e.g. coagulopathy) or thrombophilia, such as in patients with hemophilia, coagulation disorders, thrombocytopenia, etc.; Currently receiving full-dose oral or injectable anticoagulants or thrombolytic agents for therapeutic purposes (prophylactic use such as low-dose aspirin is allowed)
* Known allergies to any study drug or excipients
* Participate in other drug clinical trials within 4 weeks before randomization
* Pregnant or lactating women
* Other factors considered by the investigator to be unsuitable for participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, an average of 1 year
  Objective Response Rate
DFS | through study completion, an average of 1 year
  Disease Free Survival

SECONDARY OUTCOMES:
R0 resection rate | 1 year
  The tumor was completely removed with negative margins, meaning no residual tumor
OS | Up to 24 months
  Overall Survival
DCR | DCR will be calculated as the percentage of patients who achieved Stable Disease(SD) or better for more than 8 weeks (RECIST v1.1)
  Disease Control Rate
EFS | Up to 12/24 months
  Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Huang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No